CLINICAL TRIAL: NCT03508375
Title: Evaluation of the Serum Soluble Fractalkine as a Biomarker of Pulmonary Fibrosis in Systemic Sclerosis
Acronym: SCLEROLUNG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-03; 2018-A00066-49 (Other: N°IDRCB)
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Systemic Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SSc without ILD (Experimental)
  Interventions: Biological: blood samples
- SSc with ILD (Experimental)
  Interventions: Biological: blood samples
- patients with idiopathic pulmonary fibrosis (Active Comparator)
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — blood samples

SUMMARY:
Systemic Scleroderma (SCS) is an autoimmune disease characterized by vascular involvement, a dysimmune condition, cutaneous and visceral fibrosis. Interstitial lung disease (ILD) affects 75% of SSc patients and is the leading cause of death in SSc. No diagnostic or prognostic biomarkers of SSc-associated ILD have been validated to date. The search for such a serum biomarker is essential to assess the severity of these patients and to help the therapeutic management.

We have shown that soluble fractalkine is elevated in SSc patients, especially in SSc patients with ILD. The fractalkine is both an endothelial adhesion molecule and a chemokine that binds to the CX3CR1 receptor expressed by immune populations. It would thus reflect the vasculopathy and inflammation that lead to the fibrosing pulmonary involvement of this disease.

Objectives and means: We aim to perform a low-risk interventional biomedical research which main objective is the quantitative evaluation of soluble fractalkine in SSc patients with ILD in comparison with SSc patients without ILD. This epidemiological, explanatory, analytical, single-center study will comprise three groups: 1 / SSc without ILD (control group in the context of SSc), 2/ SSc with ILD and 3/ patients with idiopathic pulmonary fibrosis (IPF) (control group of the ILD). Secondary objectives are evaluation of: 1 / fractalkine levels in the IPF, 2 / correlations between fractalkine levels and severity of ILD and of SSc disease over time, 3 / correlations between fractalkine and 2 other biomarkers: KL-6 (marker of pulmonary fibrosis) and soluble CD146 (sCD146, marker of vasculopathy), 4 / predictive values of the decline in lung function of these 3 markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 with SSc with or without ILD with a medical follow up in AP-HM
* Patients, followed at AP-HM, with IPF

Exclusion Criteria:

* Impossibility of taking blood
* Known diagnosis of respiratory disorders other than SSc-associated ILD and IPF
* An infection in progress
* An evolutive cancer
* Chemotherapy or radiation therapy in progress
* Minors
* Pregnant or lactating women
* Majors under guardianship
* People staying in a health or social facility
* People in emergency
* Non-beneficiaries of a social security scheme
* Persons deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
fractalkine levels | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, BDR, France